CLINICAL TRIAL: NCT01501721
Title: Anthropometric and Metabolic Changes Associated With a Low-volume Home-based Exercise Program
Brief Title: Anthropometric Changes Associated With Home-based Exercise Among School Cooks
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rio de Janeiro State University (Other)
Responsible Party: Principal Investigator, Mauro Felippe Felix Mediano, Principal Investigator, Rio de Janeiro State University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: CNPq474135/2006-3
Record Dates: First submitted 2011-12-14; First posted 2011-12-29 (Estimated); Last update posted 2011-12-29 (Estimated); Status verified 2011-12

CONDITIONS: Obesity
Keywords: prevention; workers; clinical trials; obesity
MeSH Terms: conditions — Obesity | interventions — Exercise; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise (Experimental): Home-based exercise program
  Interventions: Behavioral: Exercise
- Nutritional counseling (Experimental): Nutrition counseling aiming to reduce suggar intake
  Interventions: Behavioral: Diet

INTERVENTIONS:
Behavioral: Exercise — Home-based exercise program
  Other Names: Home-based exercise group
  Arms: Exercise
Behavioral: Diet — Nutritional counseling aiming to reduce suggar intake
  Other Names: Diet group
  Arms: Nutritional counseling

SUMMARY:
Objective: This study aimed to characterize the food intake and energy expenditure of school cooks and to evaluate the anthropometric and metabolic changes that occurred after a low-volume home-based exercise program.

Methods: A randomized clinical trial in the city of Niteroi, Rio de Janeiro, Brazil, was conducted during the school year of 2007. The trial had a factorial design based on two different interventions: 1) nutritional counseling and 2) home-based exercise. The nutritional intervention was focused on decreasing the amount of sugar used in school meals by the cooks as well as decreasing their own sugar intake. The exercise program consisted of stretching and aerobic exercises that could be practiced at home, at least three times per week (40 minutes per session), with a low-to-moderate intensity.

DETAILED DESCRIPTION:
A randomized clinical trial in the city of Niteroi, Rio de Janeiro, Brazil, was conducted during the school year of 2007 (March to December 2007). The trial had a factorial design based on two different interventions: 1) nutritional counseling and 2) home-based exercise. The present study focused on the effects of exercise intervention.

Of the 36 public schools spread over five different areas, we selected 20 schools from three areas with similar demographic and socio-economic profiles. Because of the small number of male cooks (n=5), we included only women who were neither pregnant nor breastfeeding. Cooks on sick leave or those working in other capacities were excluded. A total of 101 cooks were eligible, and six refused to participate in the study.

All participants received information about the goals of the study and signed a document indicating informed consent. The study was approved by the institutional review board of the State University of Rio de Janeiro.

School cooks enrolled in the present study were public servants and work in periods of eight hours, five days per week, in three different shifts (morning, afternoon and night). They are responsible to prepare all meals served at school and cleaning up, and schools do not have any machine to help them to perform their tasks. They eat at least one meal at school.

Sample size As previously reported13), the sample size was calculated assuming an individual reduction of 10% in sugar consumption (3.4 grams) with a power of 80% and a 5% significance level. Anticipating a rate of participation agreement around 80%, the total sample size was estimated to be 80 school cooks. For this purpose, 20 schools employing a total of 130 school cooks were randomized.

Intervention Nutritional and exercise counseling were given during the school year of 2007 (eight months). The nutritional counseling group received information focused on decreasing the amount of sugar used in school meals, as well as their own sugar intake. They participated in three nutritional education meetings regarding sugar intake and food label. All activities were realized at school and required about 20 minutes. In addition, they participated in a contest to create reduced-sugar recipes and banners, and magnets promoting the reduction of sugar intake were also provided. All school cooks, from both the control and nutritional counseling groups, participated in three discussion sessions about healthy eating.

The exercise intervention group received received a booklet on physical exercises, consisted of stretching and aerobic exercises that could be practiced at home at least three times per week for 40 minutes (per session) at low-to-moderate intensity (available at www.nebin.org). The exercise sessions were divided into three parts: 1) A warm-up routine consisting of gentle body movement and stretching exercises (5 minutes); 2) An aerobic cycle performed in a circuit with continuous movements involving large arm and leg muscles, as well as exercises using a ball, ropes, stair climbing, and standing up from a chair (balls and ropes were given to the participants) (30 minutes); and 3) a cool-down period, in which the same initial stretching exercises were performed (5 minutes). The participants were encouraged to engage in exercise of low-to-moderate intensity with low impact at least three times a week during the eight months. In the first week, women were advised to perform only a 20-minute session, increasing gradually (10 minutes/session/week) up to 40 minutes per session. Each session comprised activities with balls, ropes, stairs and chair. Additionally, they were advised to reduce the exercise intensity if they felt any discomfort (e.g., if they were experiencing breathlessness or muscle aches). School cooks allocated to control group received only general information for physical activity and did not received the booklet.

Measurements The anthropometric variables were collected at three different times (baseline, 4 and 8 months), while individual food intake, based on a previously validated food frequency questionnaire14), and fasting blood samples were collected at baseline and after 8 months.

Height was measured to the nearest 0.5 cm with a wall-mounted stadiometer, and body weight was measured using the same calibrated digital scale (Tanita, BC 533 Inner Scan) for all participants. Circumference measurements were taken at the largest girth of the hip and smallest girth of the waist. All anthropometric measurements were performed according to standard techniques15).

Blood samples were collected in the morning after 10 hours of fasting. Plasma lipids and glucose were measured using GoldAnalisa kits. The LDL and VLDL cholesterol concentrations were calculated according to the Friedewald equation16) based on the triacylglycerol measurements.

Physical activity energy expenditure at baseline was evaluated in a sub-sample of 30 participants using an accelerometer (Actical® physical activity monitor, Mini Mitter, Bend, OR, USA). The accelerometer was programmed according to the manufacturer's instructions by entering the height, weight, age and sex of each subject. The subjects were instructed to place the accelerometers at their waists and wear them continuously for two consecutive days, except during activities in which contact with water could occur (e.g., during a bath).

Data analysis The characteristics of school cooks were expressed as means with standard deviations, and we compared the two intervention groups at baseline by using Student's t-test. The effects of nutritional counselling and home-based exercise on weight and circumference were evaluated through repeated random regression (RRR) analysis using PROC MIXED in SAS (version 9.1; SAS Institute Inc, Cary, NC). The analysis for the effects of exercise intervention was adjusted for dietary intervention while the analysis for the effects of nutritional counselling was adjusted for exercise intervention. The RRR is an intention-to-treat analysis because it includes all observations of each one of the subjects regardless of loss to follow-up or complies with instructions. The term of interest was treatment X time interaction, which estimates the rate of change in the outcomes over time. Residual plots of all models were examined, and their distribution did not show major deviations from regression assumptions. Changes in plasma lipids and glucose (samples of which were taken twice) between the groups were determined by Student's t-test.

ELIGIBILITY:
Inclusion Criteria:

* Of the 36 public schools spread over five different areas, we selected 20 schools from three areas with similar demographic and socio-economic profiles.

Exclusion Criteria:

* School cooks who were pregnant or breastfeeding

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2007-01; Primary Completion 2007-12 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline for weight at 4 and 8 months of follow-up | Baseline, 4 and 8 months
  Body weight was measured using the same calibrated digital scale (Tanita, BC 533 Inner Scan) for all participants

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Mediano, PhD, Principal Investigator — Rio de Janeiro State University